CLINICAL TRIAL: NCT01915680
Title: Intraocular Pressure Fluctuation in Patients With Glaucoma and in Healthy Patients During Standard Yoga Positions
Status: Completed | Type: Observational
Sponsor: Robert Ritch, MD, LLC. (Other)
Responsible Party: Principal Investigator, Robert Ritch, MD, Associate Professor of Ophtalmology, Robert Ritch, MD, LLC.
Other Study IDs: NYGRI Yoga Study 13.04
Record Dates: First submitted 2013-07-12; First posted 2013-08-05 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2013-12

CONDITIONS: Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma
- Control

SUMMARY:
The purpose of the study is to investigate the IOP difference between normal and glaucomatous eyes using standard ophthalmic tonometry devices while subjects are performing different standard yoga asanas. The IOP of participants will be measured prior, immediately at start of the asana, 2 minutes into the asana, and immediately after assuming a sitting position. The patient will wait 10 minutes and a final IOP will be taken. Four standard yoga asanas will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma or healthy control
* Practice yoga
* 18-80 years old
* Practice Yoga for a minimum of 12 months

Exclusion Criteria:

* Healthy subjects do not have normal ophthalmic exam
* Cannot maintain yoga positions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma Practice and Yoga Studios
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure | Change from Baseline, Immediate, 2 Minutes, Post, 10 min Post

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States

REFERENCES:
- [Derived] Jasien JV, Jonas JB, de Moraes CG, Ritch R. Intraocular Pressure Rise in Subjects with and without Glaucoma during Four Common Yoga Positions. PLoS One. 2015 Dec 23;10(12):e0144505. doi: 10.1371/journal.pone.0144505. eCollection 2015. PMID 26698309